CLINICAL TRIAL: NCT06246110
Title: A Phase 2 Study of EIK1001 in Combination With Pembrolizumab and Chemotherapy in Patients With Stage 4 Non-Small Cell Lung Cancer
Brief Title: A Phase 2 Study of EIK1001 in Combo With Pembrolizumab and Chemotherapy in Patients With Stage 4 NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eikon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EIK1001-005
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: NSCLC
Keywords: Squamous; Nonsquamous; Metastatic
MeSH Terms: conditions — Neoplasm Metastasis | interventions — pembrolizumab; Paclitaxel; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A - Participants with non-squamous NSCLC (Experimental): Participants in this arm will receive EIK1001 + Standard of Care (SOC).
  Interventions: Drug: EIK1001; Drug: Pembrolizumab; Drug: Pemetrexed; Drug: Carboplatin
- Cohort B - Participants with squamous NSCLC (Experimental): Participants in this arm will receive EIK1001 + Standard of Care (SOC).
  Interventions: Drug: EIK1001; Drug: Pembrolizumab; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: EIK1001 — EIK1001 is a Toll like receptor 7/8 (TLR 7/8) agonist
Drug: Pembrolizumab — PD-1 inhibitor
Drug: Paclitaxel — Chemotherapy
  Arms: Cohort B - Participants with squamous NSCLC
Drug: Pemetrexed — Chemotherapy
  Arms: Cohort A - Participants with non-squamous NSCLC
Drug: Carboplatin — Chemotherapy

SUMMARY:
This study is for patients with advanced/metastatic non-small cells lung cancer (NSCLC) who have not received any treatment through the vein for the advanced disease.

DETAILED DESCRIPTION:
This is a multicenter open-label phase 2 trial that aim to assess the safety, tolerability, and efficacy of EIK1001 in combination with standard of care in participants with both confirmed stage 4 squamous and non-squamous NSCLC who have not received prior systemic therapy for the advanced disease. The study includes dose finding and evaluates adverse events and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. be ≥ 18 years of age on the day of signing of informed consent.
2. confirmed Stage 4 NSCLC (squamous or non-squamous) and be considered for standard of care.
3. have confirmation that mutation-directed therapy is not indicated (documentation of absence of tumor activating mutations/fusions that are approved for first line therapy).
4. have at least 1 lesion with measurable disease at Baseline according to RECIST 1.1 as determined by the local site Investigator/radiology assessment.
5. have not received prior systemic treatment for advanced/metastatic NSCLC.
6. have an ECOG Performance Status of 0 to 1.
7. have adequate organ function.

Exclusion Criteria:

1. does not have predominantly squamous cell or non-squamous cell histology NSCLC. Mixed tumors will be categorized by the predominant cell type; if small cell elements are present, the participant is ineligible.
2. is currently participating in or has participated in a study of an investigational agent and received investigational therapy within 4 weeks or 5 half-lives (whichever is shorter) of administration of EIK1001.
3. prior to the first dose of EIK1001, has received prior systemic therapy for metastatic disease, or had major surgery (< 3 weeks prior to the first dose).
4. has completed palliative radiotherapy within 7 days of the first dose of study drug administration.
5. has a known history of prior malignancy, except if the participant has undergone potentially curative therapy with no evidence of that disease recurrence for 5 years.
6. has an active infection requiring therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with safety event during treatment | Up to 2 years
  Defined AEs that occur during treatment and are deemed to be related EIK1001 or combination with SOC or due to disease progression or toxicity.

SECONDARY OUTCOMES:
Percentage of participants with objective response rate (ORR) and duration of response (DOR). | Up to 4 years
  Objective response (OR) is defined as participants who have a confirmed complete response (CR) or partial response (PR) by RECIST 1.1 and DOR is defined as the time from the first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first, in participants demonstrating CR or PR, as assessed by the investigator.

OTHER OUTCOMES:
Overall Survival (OS) at Final Follow-Up | Up to 4 years
  OS defined as the time from the first dose of study medication to death due to any cause
Progression Free Survival (PFS) | Up to 4 years
  Progression-free survival (PFS) is defined as the time from the first dose of the study medication to the first documented disease progression by RECIST 1.1 (Investigator) or death due to any cause, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Etah Kurland, MD, Study Director — Eikon Therapeutics
Locations (39):
- United States (39):
  - Southern Cancer Care, Daphne, Alabama
  - Ironwood Cancer and Research Center, Chandler, Arizona
  - California Cancer Care Associates for Research & Excellence, Fresno, California
  - California Research Institute, Los Angeles, California
  - University of Southern California, Norris Comprehensive Cancer Center, Los Angeles, California
  - Providence St Joseph Hospital, Center for Cancer Prevention and Treatment, Orange, California
  - Sutter Health Institute for Medical Research, Sacramento, California
  - Rocky Mountain Cancer, Lone Tree, Colorado
  - Bioresearch Partner, Hialeah, Florida
  - Memorial Cancer Institute, Hollywood, Florida
  - Mid-Florida Hematology and Oncology Center, Orange, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Atlanta Piedmont Hospital, Atlanta, Georgia
  - Kaiser Permanente Hawaii, Honolulu, Hawaii
  - Illinois Cancer Specialists, Niles, Illinois
  - Accelacare of Duly, Tinley Park, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Health Midwest Oncology Associates of Kansas, Overland Park, Kansas
  - Cancer Center of Kansas, Wichita, Kansas
  - Medstar Franklin Square Cancer Center at Loch Raven Campus, Baltimore, Maryland
  - Maryland Oncology, Columbia, Maryland
  - Jersey Shore University Medical Center/Meridian Hematology & Oncology, Neptune City, New Jersey
  - New York Cancer and Blood Specialists, Babylon, New York
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Weil Cornell Medical Center, New York, New York
  - Albert Einstein College of Medicine, Jacobi Medical Center, The Bronx, New York
  - Cancer and Blood Specialists of New York, White Plains Hospital, White Plains, New York
  - Messino Cancer Centers, Asheville, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Willamette Valley, Eugene, Oregon
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - Baptist Cancer Center, Memphis, Tennessee
  - Texas Oncology, Austin, Austin, Texas
  - Texas Oncology, Bedford, Bedford, Texas
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Blue Ridge Cancer Care Oncology Associates SW VA, Blacksburg, Virginia
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Shenandoah Oncology, Winchester, Virginia